CLINICAL TRIAL: NCT03373201
Title: Evaluating the Effects of Tasimelteon vs. Placebo on Jet Lag Type Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VEC-162-3107
Record Dates: First submitted 2017-10-31; First posted 2017-12-14 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Jet Lag Type Insomnia
MeSH Terms: interventions — tasimelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tasimelteon (Experimental)
  Interventions: Drug: Tasimelteon
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tasimelteon — Oral capsule
  Arms: Tasimelteon
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate tasimelteon vs. placebo on sleep in healthy individuals after a phase advance in jet lag type insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Ability and acceptance to provide written consent, fluent in English;
* Healthy subjects with no medical, psychiatric or current sleep disorders;
* Men or women between 18-75 years;
* Body Mass Index of ≥ 18 and ≤ 30 kg/m2.

Exclusion Criteria:

* Major surgery, trauma, illness or immobile for 3 or more days within the past month;
* Pregnancy or recent pregnancy (within 6 weeks);
* A positive test for drugs of abuse at the screening or evaluation visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Vanda Investigational Site, Little Rock, Arkansas
  - Vanda Investigational Site, Alameda, California
  - Vanda Investigational Site, San Diego, California
  - Vanda Investigational Site, Santa Monica, California
  - Vanda Investigational Site, Oakland Park, Florida
  - Vanda Investigational Site, Atlanta, Georgia
  - Vanda Investigational Site, Chevy Chase, Maryland
  - Vanda Investigational Site, St Louis, Missouri
  - Vanda Investigational Site, New York, New York
  - Vanda Investigational Site, Cincinnati, Ohio
  - Vanda Investigational Site, Oklahoma City, Oklahoma
  - Vanda Investigational Site, Houston, Texas

REFERENCES:
- [Derived] Polymeropoulos CM, Mohrman MA, Keefe MS, Brzezynski JL, Wang J, Prokosch LS, Polymeropoulos VM, Xiao C, Birznieks G, Polymeropoulos MH. Efficacy of Tasimelteon (HETLIOZ(R)) in the Treatment of Jet Lag Disorder Evaluated in an 8-h Phase Advance Model; a Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial. Front Neurol. 2020 Jul 9;11:611. doi: 10.3389/fneur.2020.00611. eCollection 2020. PMID 32754110

RESULTS

PARTICIPANT FLOW:
Groups:
- Tasimelteon: 20 mg tasimelteon capsule PO Daily, 1 Day
- Placebo: Placebo capsule PO Daily, 1 Day
Period: Overall Study
Arm/Group | Tasimelteon | Placebo
Started | 160 | 160
Completed | 159 | 159
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tasimelteon | Placebo | Total
Number analyzed (Participants) | 159 | 159 | 318
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (11.20) | 35.9 (12.63) | 35.8 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 81 | 167
  Male | 73 | 78 | 151
Race/Ethnicity, Customized [Number; unit: participants]
  White | 94 | 97 | 191
  Black or African American | 44 | 47 | 91
  Asian | 15 | 13 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time in the First Two Thirds of the Night
Description: Total sleep time during the first 2/3 of the night following an 8-hour phase advance bedtime, as measured by PSG. This is representative of trans meridian travel across 8 time zones.
Time Frame: 1 Day
Population: Intent-to-Treat Population
Measure: Least Squares Mean (Standard Deviation); unit: Minutes
Groups:
- Tasimelteon: Tasimelteon: 20mg Oral Capsule
Arm/Group | Placebo | Tasimelteon
Number analyzed (Participants) | 159 | 159
Minutes | 156.1 (80.67) | 216.4 (69.69)
Statistical Analysis 1: Comparison: Placebo vs Tasimelteon; Test type: Superiority; p < .0001, ANOVA; Difference between LS means = 60.3, 95% CI 2-sided [44.0 to 76.7]

2. Secondary Outcome: Total Sleep Time
Description: Total Sleep Time as measured by PSG.
Time Frame: 1 Day
Population: Intent-to-Treat Population
Measure: Least Squares Mean (Standard Deviation); unit: Minutes
Groups:
- Tasimelteon: Tasimelteon: 20 mg Oral Capsule
Arm/Group | Placebo | Tasimelteon
Number analyzed (Participants) | 159 | 159
Minutes | 230.3 (97.39) | 315.8 (95.51)
Statistical Analysis 1: Comparison: Placebo vs Tasimelteon; Test type: Superiority; p < .0001, ANOVA; Difference between LS Means. = 85.5, 95.0% CI 2-sided [64.3 to 106.6]

3. Secondary Outcome: Latency to Persistent Sleep
Description: Length of time elapsed between lights out and onset of persistent sleep as measure by PSG.
Time Frame: 1 Day
Population: Intent-to-Treat Population
Measure: Least Squares Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | Tasimelteon
Number analyzed (Participants) | 159 | 159
Minutes | 36.8 (63.56) | 21.8 (33.69)
Statistical Analysis 1: Comparison: Placebo vs Tasimelteon; Test type: Superiority; p < .0001, ANOVA; Difference between LS means = -15.1, 95% CI 2-sided [-26.2 to -4.0]

4. Secondary Outcome: Wake After Sleep Onset
Description: The amount of wake time during the sleep period after sleep onset (as measured by polysomnography).
Time Frame: 1 Day
Population: Intent-to-Treat Population
Measure: Least Squares Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | Tasimelteon
Number analyzed (Participants) | 159 | 159
Minutes | 219.1 (96.90) | 144.6 (86.73)
Statistical Analysis 1: Comparison: Placebo vs Tasimelteon; Test type: Superiority; p < .0001, ANOVA; Difference between LS means = -74.6, 95% CI 2-sided [-94.8 to -54.3]

5. Secondary Outcome: Next Day Alertness as Measured by the Karolinska Sleepiness Scale (Night 1 Average Score)
Description: A 9-point scale that measures subjective levels of fatigue by asking how sleepy subjects feel at that moment: 1 = extremely awake to 9 =extremely sleepy/fighting to stay awake.
Time Frame: 1 Day
Population: Intent-to-Treat Population
Measure: Least Squares Mean (Standard Deviation); unit: Night 1 average score
Arm/Group | Placebo | Tasimelteon
Number analyzed (Participants) | 159 | 159
Night 1 average score | 4.5 (1.86) | 4.0 (1.77)
Statistical Analysis 1: Comparison: Placebo vs Tasimelteon; Test type: Superiority; p = 0.0083, ANOVA; Difference between LS Means. = -0.5, 95.0% CI 2-sided [-0.9 to -0.1]

6. Secondary Outcome: Next Day Alertness as Measured by the Visual Analogue Scale (Night 1 Average Score)
Description: The VAS was a self-rated scale to assess sleepiness. Participants marked along a 100 mm line to represent their current state of sleepiness, 0 being very sleepy and 100 being very alert. The VAS was administered four times following the dose administration after awakening.
Time Frame: 1 Day
Population: Intent-to-Treat Population
Measure: Least Squares Mean (Standard Deviation); unit: Night 1 Average Score in millimeters
Arm/Group | Placebo | Tasimelteon
Number analyzed (Participants) | 159 | 159
Night 1 Average Score in millimeters | 54.2 (23.46) | 60.8 (22.24)
Statistical Analysis 1: Comparison: Placebo vs Tasimelteon; Test type: Superiority; p = 0.0099, ANOVA; Difference between LS Means. = 6.6, 95.0% CI 2-sided [1.6 to 11.6]

ADVERSE EVENTS:
Time Frame: AE Data collected over the 1 Day/ 1 Night study plus a 30 day follow up period
Arm/Group | Tasimelteon | Placebo
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/160
Serious Adverse Events (participants affected / at risk) | 1/160 | 0/160
Other Adverse Events (participants affected / at risk) | 8/160 | 4/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tasimelteon (N=160) | Placebo (N=160)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — There was only one serious adverse event of atrial fibrillation in a subject receiving tasimelteon that was assessed as unrelated to study treatment and related to previously undiagnosed hyperthyroidism.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tasimelteon (N=160) | Placebo (N=160)
Headache (Nervous system disorders) | 8 (8) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT03373201/Prot_SAP_001.pdf